CLINICAL TRIAL: NCT03642639
Title: A Prospective, Multi-center, Single Arm Study to Obtain "Real World" Clinical Data and Characterize the Acute and Long-term Performance of the MICRUSFRAME and GALAXY Coils Including the PulseRider Aneurysm Neck Reconstruction Device for the Endovascular Treatment of Intracranial Aneurysms
Brief Title: A Study to Look at Performance of MICRUSFRAME and GALAXY Coils for the Treatment of Intracranial Aneurysms
Acronym: STERLING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cerenovus, Part of DePuy Synthes Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNV_2017_01
Record Dates: First submitted 2018-07-11; First posted 2018-08-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Aneurysms
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Coils (Other): MICRUSFRAME and GALAXY coils
  Interventions: Device: MICRUSFRAME and GALAXY coils

INTERVENTIONS:
Device: MICRUSFRAME and GALAXY coils — MICRUSFRAME and GALAXY Coils

SUMMARY:
A post-market registry evaluating ruptured/unruptured aneurysms treated with MICRUSFRAME and GALAXY coils

DETAILED DESCRIPTION:
A registry to collect real world data on the use of Cerenovus coils. The study will be a post-market registry evaluating ruptured/unruptured aneurysms treated with MICRUSFRAME and GALAXY coils

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 21 and 80 years of age
2. Patient has an intracranial saccular aneurysm, ruptured or unruptured, suitable for embolization with coils
3. Patient is able and willing to comply with protocol and follow-up requirements

Exclusion Criteria:

1. Pre-planned staged procedure on unruptured aneurysm
2. More than one aneurysm requiring treatment during the course of study
3. Fusiform aneurysm

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 809 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Occlusion Rate | 12 Months
  Occlusion rate at 12 Months post procedure

SECONDARY OUTCOMES:
1. Packing Density | From enrollment to end of treatment at 12 months
  Packing density will be evaluated based on aneurysm volume and the coils used during the procedure.
2. Complete occlusion rate | 12 month
  Complete occlusion rate at 12 month follow-up
3. Recanalization Rate | 12 Months
  Recanalization Rate: Any worsening of occlusion grading at 12 Month follow-up
4. Device related serious adverse events | 12 Months
  Any device related serious adverse events will be reported through 12 month follow-up
5. Retreatment Rate | 12 Months
  Aneurysm re-treatment rates will be tracked and recorded during the 12 month follow-up
6. Modified Rankin Score | 12 Months
  Modified Rankin Score (Scale from 0-6) at 12 Months. 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
7. Length of hospital stay | From enrollment to 12 Months
  Hospital stay length will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Reade De Leacy, Principal Investigator — Mount Sinai Hospital, New York; Osama Zaidat, Principal Investigator — Mercy Health St. Vincent Hospital
Locations (51):
- United States (30):
  - University of Arizona, Tucson, Arizona
  - Mercy San Juan Medical Center, Carmichael, California
  - University of California Irvine, Orange, California
  - University of Florida, Gainesville, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Memorial Health University, Savannah, Georgia
  - Rush University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Javon Bea Hospital, Rockford, Illinois
  - Norton Healthcare, Louisville, Kentucky
  - Maine Medical Center, Scarborough, Maine
  - University of Massachusetts, Worcester, Massachusetts
  - St. Louis University, St Louis, Missouri
  - University of Buffalo, Buffalo, New York
  - Mount Sinai Hospital, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Westchester Medical Center, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Mercy Health St. Vincent Medical Center, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Clinic, Danville, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Tennessee Interventional and Imaging Associates, Chattanooga, Tennessee
  - University of Tennessee, Knoxville, Tennessee
  - Texas Stroke Institute, Plano, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
- Algemeen Ziekenhuis Groeninge, Kortrijk, Belgium
- France (5):
  - Centre Hospitalier Universitaire d'Amiens Picardie, Amiens
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Hopital Roger Salengro-Centre Hospitalier Universitaire de Lille, Lille
  - Praticien Hospitalier Université de Lorraine, Nancy
  - Centre Hospitalier Regional Universitaire de Tours, Tours
- Universitatsklinikum Schleswig Holstein, Lübeck, Germany
- Galilee Hospital Naharyia, Nahariya, Israel
- Italy (3):
  - Ospedale Niguarda Ca' Granda, Milan
  - Policlinico Tor Vergata, Roma
  - Ospedale Cannizzaro, Sicily
- Japan (6):
  - Aichi Medical University Hospital, Aichi
  - Okayama University Hospital, Okayama
  - National Hospital Organization Osaka National Hospital, Osaka
  - Tominaga Hospital, Osaka
  - Kohnan Hospital, Sendai
  - Meihokai Yokohama Shin-Toshi Brain Orthopedic Hospital, Yokohama
- Centro Hospitalar de Vila Nova de Gaia, Porto, Portugal
- Hospital Universitari i Politecnic La Fe, Valencia, Spain
- Switzerland (2):
  - Hopitaux Universitaires de Geneve, Geneva
  - University Hospital Zurich, Zurich